CLINICAL TRIAL: NCT06650618
Title: Twelve Leads Electrocardiographic Expressions at Different Body Positioning
Status: Not yet recruiting | Type: Observational
Sponsor: Kaohsiung Medical University Chung-Ho Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: KMUHIRB-E(I)-20240272
Record Dates: First submitted 2024-09-25; First posted 2024-10-21 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-08

CONDITIONS: Electrocardiogram
Keywords: ECG; heart rhythm; electrical conduction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Electrical conduction in the heart produces a heartbeat; electrical signals are sent to the heart muscle upon each contraction, causing the heart to pump blood. These electrical impulses are recorded by an electrocardiogram (ECG), which makes it possible to evaluate electrical conduction and cardiac rhythm. ECG is a non-invasive technique used to assess pacemaker function and perioperative heart health. Ten electrodes are used in the 12-lead ECG, the gold standard for diagnosing cardiac illness and anatomy, to record the electrical activity of the heart from various perspectives. With wireless data transmission to the cloud, this technology is now included into emergency and ambulance situations, streamlining processes and improving signal quality. The purpose of this observational study is to examine 12-lead electrocardiogram data for better clinical application and diagnosis.

DETAILED DESCRIPTION:
The heartbeat is a result of electrical conduction in the heart. The heart's contractions release electrical signals that trigger the heart muscle to pump blood to the lungs and the rest of the body. An electrocardiogram (ECG) records these electrical signals from each heartbeat, allowing for the observation of heart rhythm and the assessment of any abnormalities in electrical conduction. The ECG is a non-invasive monitoring tool used for evaluating heart health throughout the perioperative period and for checking the function of pacemakers. By analyzing the shape, size, and time intervals of these waveforms, ECGs provide visual representations that help healthcare professionals assess conditions related to heart valve diseases.

The 12-lead ECG is considered the gold standard for evaluating cardiac structure and diagnosing various heart conditions. This system consists of twelve leads created from ten electrodes, recording the heart rates electrical activity from different angles in three-dimensional space to understand the condition of various heart regions. Currently, 12-lead ECG machines are widely used in emergency and ambulance settings. They often incorporate integrated electrode patches that replace the traditional ten individual electrode patches, significantly simplifying the process and reducing errors. This integration improves signal transmission and quality compared to traditional ECG leads. Data is transmitted wirelessly, paired with mobile device software, and sent to the cloud to support diagnostic reports.

This study is an observational research project aimed at establishing and analyzing 12-lead ECG data. The goal is to utilize this data for more in-depth diagnostics and to observe its differences and clinical applications.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18~65 years of age
* Fluent in either Taiwanese/Chinese/English.

Exclusion Criteria:

* Pregnancy
* Refusal to give informed consent
* Candidate for coronary bypass surgery or valves surgery or other cardiac surgery
* Participants with diagnosed arrhythmia, ischemic heart disease or congestive heart failure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants without diagnosed arrhythmia, ischemic heart disease, congestive heart failure or pending for all kinds of heart surgery.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-10-31 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
ECG change related to position | through study completion, an average of 30 minutes.
  ECG ST segment elevation or depression might be attributed to varying body postures. The ST segments' change to baseline will be compared by the investigators.

CONTACTS AND LOCATIONS:
Overall Officials: Tzu-Ying Li, Study Director — Kaohsiung Medical University Chung-Ho Memorial Hospital
Locations (1):
- Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City, Sanmin Dist, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Statistical Analysis Plan can be shared
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months and ending 1 year after the publication of results
Access Criteria: Researchers with formal inquiry will be able to access it.